CLINICAL TRIAL: NCT04311385
Title: Management and Evolution of Acute Diverticulitis With Pericolic Free Gas - a Multicentre Observational Study
Brief Title: Management and Evolution of Acute Diverticulitis With Pericolic Free Gas
Acronym: ADiFas
Status: Completed | Type: Observational
Sponsor: Hospital Central de la Defensa Gómez Ulla (Other)
Responsible Party: Principal Investigator, Patricia Tejedor, Colorectal Consultant Surgeon, Hospital Central de la Defensa Gómez Ulla
Other Study IDs: 8_20
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Diverticulitis; Diverticulitis Colon; Diverticulitis; Perforation, Bowel; Diverticulitis of Sigmoid
Keywords: Acute diverticulitis; Hinchey; Management of diverticulitis; Treatment of diverticulitis; Diverticulitis classification
MeSH Terms: conditions — Diverticulitis; Diverticulitis, Colonic | interventions — Postmortem Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diverticulitis: Patients admitted as an emergency with acute diverticulitis diagnosed by CT scan.
  Inclusion criteria
  * Patients over 18 years old
  * Informed consent form signed
  * Diagnosed of acute diverticulitis
  * CT scan reported as 1-2 pericolic bubbles with or without free fluid
  Exclusion criteria
  o CT scan showing free distant bubbles in the abdomen
  Interventions: Diagnostic Test: CT imaging

INTERVENTIONS:
Diagnostic Test: CT imaging — CT scan reported as 1-2 pericolic bubbles, but no free distant bubbles in the abdomen or abscess.

SUMMARY:
The severity of diverticulitis is usually graded with the use of modified Hinchey Criteria. However, there is a condition often seen in the CT scan that is not included in this classification itself; 1-2 pericolic bubbles but no free air or fluid into the abdomen or above the liver. Outcome in these patients remains unknown. We aim to analyse the treatment that these patients and their evolution over the first year after the diagnosis in order to predict the disease related outcome.

The study is set up as a retrospective multicentre observational study. Inclusion criteria are Patients over 18 years old, Diagnosed of acute diverticulitis with a CT scan reported as 1-2 pericolic bubbles with or without free fluid. Exclusion criteria: 1) CT scan showing free distant bubbles in the abdomen. 2) CT scan showing abscess.

Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a two-sided test, 137 subjects are necessary in the observed group to recognize a difference in morbidity greater than or equal to 10%. A proportion in the reference group has been estimated to be 20%. It has been anticipated a drop-out rate of 0%.

Primary outcome is 30-day morbidity and mortality. Secondary outcomes include malignancy and 1 year morbidity including recurrences and ongoing disease. Data will be collected in an online repository. The CT scans will be reviewed by 2 experienced independent radiologists. The management of these patients at the moment of the diagnosis will be recorded, as well as their evolution over the first year during the outpatient clinics. Figure 1 represents the study flow chart.

Data will be collected in an online secure and protected repository (Castor edc). The planned study period is 2 years (01/06/2020 - 31/12/2021).

CT scans will be reviewed by 2 experienced radiologists. Every other CT scan performed during the follow-up will be reviewed by the same radiologists.

The management of these patients at the moment of the diagnosis will be recorded, as well as their evolution over the first year during the outpatient clinics.

This study protocol is a new approach to an unknown entity in diverticulitis. We are convince that the outcomes are clinically relevant to patients and interesting for all physicians treating diverticulitis.

DETAILED DESCRIPTION:
Diverticular disease of the colon is a common disease that includes diverticulosis and diverticulitis. Most patients who have diverticulosis remain asymptomatic; however an estimated 15-20% will develop acute diverticulitis (AD).(1) AD is an inflammatory condition affecting at least one colonic diverticula, often associated with pericolonic inflammation.(2) Diverticulitis can range form mild to severe. Severe, complicated cases with perforation may be associated with intra-abdominal abscess, generalized, purulent peritonitis, fistula formation, bleeding or obstruction. The extent of the perforation determines the clinical behavior. Microperforations remain localised because they are contained by pericolic fat and mesentery, leading to the formation of small pericolic abscesses.

The gold standard for the diagnosis of diverticulitis is the Computed Tomography (CT). It has a sensitivity ranging form 85% to 97% (3,4) and it is very accurate identifying colonic perforation, which can have a direct impact on the management of the patient. The severity of diverticulitis is usually graded with the use of modified Hinchey's Criteria, based on CT imaging and on preoperative findings.(5) It distinguishes four stages of acute complicated diverticulitis. Several modifications to the Hinchey classification have been proposed due to the advancements in imaging modalities. New subcategories have been added that take radiological findings into consideration.(6) However, there is a condition often seen in the CT scan that is not included in this classification itself; a single pericolic bubble.

The management of AD depends on its severity and complexity, and it requires hospitalization, bowel rest and surgery in selected cases. Antibiotic therapy is part of the management of complicated diverticulitis and recent guidelines are in accordance at recommending broad-spectrum antibiotics. Biondo and colleagues evaluated 92 papers in a systematic review, concluding that patients with severe AD without need of emergency surgery, should be treated with hospitalization, parenteral fluids and a single intravenous antibiotic active against aerobic and anaerobic bacteria.(7) Approximately 15-20% of patients admitted with AD have an abscess on CT scan.(8) The size of 3-6 cm has been generally accepted to be treated with antibiotics vs. percutaneous drainage.(8-10) However, clinical monitoring is mandatory and a CT scan should be repeated if the patient does not show clinical and laboratory improvement.

In the 1990s laparoscopic lavage (LL) was proposed to treat patients affected by peritonitis due to perforated AD.(11) Initial results encouraged surgeons to perform LL;(12-14) however, in the 2000s three Randomized Control Trials (RCT) were published with mixed results.(15-17) Two of them suggested that the traditional surgical treatment (segmental resection and stoma formation) achieves more successful results.(16,17) In summary, there are several guidelines for the treatment of AD regarding its severity; however, there is no consensus in the management of those patients with 1-2 pericolic bubbles but no free air into the abdomen. The treatment that these patients receive is widely variable.

For this reason, patients admitted in the emergency unit and diagnosed of acute diverticulitis with a free pericolic bubble of air, regardless the Hinchey's criteria assigned and the treatment received, would be included in this study. We aim to analyse the treatment that they underwent and the evolution of these patients over the first year after the diagnosis. The patients will not undergo any treatment or test that would not be necessary during their follow-up out of this observational and retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Informed consent
* Diagnosed of acute diverticulitis
* CT scan reported as 1-2 pericolic bubbles with or without free fluid.

Exclusion Criteria:

* CT scan showing free distant bubbles in the abdomen
* CT scan showing abscess

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Emergency unit Hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
30-day morbidity | 30 days
  * Diverticulitis recurrence
  * Perforation (with purulent/fecal peritonitis)
  * Fistula
  * Symptomatic colonic stenosis
  * Intraabdominal abcess
  * Stoma formation
  * Emergency surgery or re-operation
  * Peri- and postoperative complications (Dindo-Clavien classification)

SECONDARY OUTCOMES:
30-day mortality | 30 days
  Death within 30 days
Malignancy | 60 days
  Malignancy in the pathological report in cases undergoing surgery
1-year morbidity | 1 year
  * Diverticulitis recurrence
  * Perforation (with purulent/fecal peritonitis)
  * Fistula
  * Symptomatic colonic stenosis
  * Intraabdominal abcess
  * Stoma formation
  * Emergency surgery or re-operation
  * Peri- and postoperative complications (Dindo-Clavien classification)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Tejedor, Consultant, Principal Investigator — Hospital Central de la Defensa Gómez Ulla
Locations (1):
- Hospital Central de la Defensa Gómez Ulla, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR)

REFERENCES:
- [Result] Kaiser AM, Jiang JK, Lake JP, Ault G, Artinyan A, Gonzalez-Ruiz C, Essani R, Beart RW Jr. The management of complicated diverticulitis and the role of computed tomography. Am J Gastroenterol. 2005 Apr;100(4):910-7. doi: 10.1111/j.1572-0241.2005.41154.x. PMID 15784040
- [Result] Jacobs DO. Clinical practice. Diverticulitis. N Engl J Med. 2007 Nov 15;357(20):2057-66. doi: 10.1056/NEJMcp073228. No abstract available. PMID 18003962
- [Result] Halligan S, Saunders B. Imaging diverticular disease. Best Pract Res Clin Gastroenterol. 2002 Aug;16(4):595-610. doi: 10.1053/bega.2002.0323. PMID 12406453
- [Result] Farrell RJ, Farrell JJ, Morrin MM. Diverticular disease in the elderly. Gastroenterol Clin North Am. 2001 Jun;30(2):475-96. doi: 10.1016/s0889-8553(05)70191-6. PMID 11432301
- [Result] Wasvary H, Turfah F, Kadro O, Beauregard W. Same hospitalization resection for acute diverticulitis. Am Surg. 1999 Jul;65(7):632-5; discussion 636. PMID 10399971
- [Result] Biondo S, Lopez Borao J, Millan M, Kreisler E, Jaurrieta E. Current status of the treatment of acute colonic diverticulitis: a systematic review. Colorectal Dis. 2012 Jan;14(1):e1-e11. doi: 10.1111/j.1463-1318.2011.02766.x. PMID 21848896
- [Result] Andersen JC, Bundgaard L, Elbrond H, Laurberg S, Walker LR, Stovring J; Danish Surgical Society. Danish national guidelines for treatment of diverticular disease. Dan Med J. 2012 May;59(5):C4453. PMID 22549495
- [Result] Ambrosetti P, Chautems R, Soravia C, Peiris-Waser N, Terrier F. Long-term outcome of mesocolic and pelvic diverticular abscesses of the left colon: a prospective study of 73 cases. Dis Colon Rectum. 2005 Apr;48(4):787-91. doi: 10.1007/s10350-004-0853-z. PMID 15747071
- [Result] Brandt D, Gervaz P, Durmishi Y, Platon A, Morel P, Poletti PA. Percutaneous CT scan-guided drainage vs. antibiotherapy alone for Hinchey II diverticulitis: a case-control study. Dis Colon Rectum. 2006 Oct;49(10):1533-8. doi: 10.1007/s10350-006-0613-3. PMID 16988856
- [Result] O'Sullivan GC, Murphy D, O'Brien MG, Ireland A. Laparoscopic management of generalized peritonitis due to perforated colonic diverticula. Am J Surg. 1996 Apr;171(4):432-4. doi: 10.1016/S0002-9610(97)89625-0. PMID 8604837
- [Result] Sorrentino M, Brizzolari M, Scarpa E, Malisan D, Bruschi F, Bertozzi S, Bernardi S, Petri R. Laparoscopic peritoneal lavage for perforated colonic diverticulitis: a definitive treatment? Retrospective analysis of 63 cases. Tech Coloproctol. 2015 Feb;19(2):105-10. doi: 10.1007/s10151-014-1258-1. Epub 2014 Dec 31. PMID 25550116
- [Result] Myers E, Hurley M, O'Sullivan GC, Kavanagh D, Wilson I, Winter DC. Laparoscopic peritoneal lavage for generalized peritonitis due to perforated diverticulitis. Br J Surg. 2008 Jan;95(1):97-101. doi: 10.1002/bjs.6024. PMID 18076019
- [Result] Taylor CJ, Layani L, Ghusn MA, White SI. Perforated diverticulitis managed by laparoscopic lavage. ANZ J Surg. 2006 Nov;76(11):962-5. doi: 10.1111/j.1445-2197.2006.03908.x. PMID 17054542
- [Result] Angenete E, Thornell A, Burcharth J, Pommergaard HC, Skullman S, Bisgaard T, Jess P, Lackberg Z, Matthiessen P, Heath J, Rosenberg J, Haglind E. Laparoscopic Lavage Is Feasible and Safe for the Treatment of Perforated Diverticulitis With Purulent Peritonitis: The First Results From the Randomized Controlled Trial DILALA. Ann Surg. 2016 Jan;263(1):117-22. doi: 10.1097/SLA.0000000000001061. PMID 25489672
- [Result] Schultz JK, Yaqub S, Wallon C, Blecic L, Forsmo HM, Folkesson J, Buchwald P, Korner H, Dahl FA, Oresland T; SCANDIV Study Group. Laparoscopic Lavage vs Primary Resection for Acute Perforated Diverticulitis: The SCANDIV Randomized Clinical Trial. JAMA. 2015 Oct 6;314(13):1364-75. doi: 10.1001/jama.2015.12076. PMID 26441181
- [Result] Vennix S, Musters GD, Mulder IM, Swank HA, Consten EC, Belgers EH, van Geloven AA, Gerhards MF, Govaert MJ, van Grevenstein WM, Hoofwijk AG, Kruyt PM, Nienhuijs SW, Boermeester MA, Vermeulen J, van Dieren S, Lange JF, Bemelman WA; Ladies trial colloborators. Laparoscopic peritoneal lavage or sigmoidectomy for perforated diverticulitis with purulent peritonitis: a multicentre, parallel-group, randomised, open-label trial. Lancet. 2015 Sep 26;386(10000):1269-1277. doi: 10.1016/S0140-6736(15)61168-0. Epub 2015 Jul 22. PMID 26209030
- [Derived] Tejedor P, Pastor C, Pellino G, Di Saverio S, Gorter-Stam M, Sylla P, Francis N; Collaborative Study Group. Management of acute diverticulitis with pericolic free gas (ADIFAS): an international multicenter observational study. Int J Surg. 2023 Apr 1;109(4):689-697. doi: 10.1097/JS9.0000000000000213. PMID 37010145